CLINICAL TRIAL: NCT04492098
Title: Analysis of Mucosal-Associated Invariant T (MAIT) Cells in Cases of Spontaneous and Recurrent Miscarriage
Brief Title: Mucosal-Associated Invariant T Cells in Cases of Miscarriage
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: MAIT-RPL
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: women with spontaneous miscarriage
  Interventions: Diagnostic Test: MAIT cells

INTERVENTIONS:
Diagnostic Test: MAIT cells — 1- Decidual tissues will be washed in phosphate buffer saline (PBS), and then preserved in Rosewell Park Memorial Institute (RPMI) 1640 medium supplemented with 100 U/mL penicillin, 100 mg/mL streptomycin and 5% fetal bovine serum (GIBCO BRL, Thermo Fisher Scientific, USA) until transfer to the laboratory. At the flow cytometry laboratory, the tissue samples will be minced finely and enzymatically digested by adding 3 ml collagenase enzyme type Ia and 2 ml PBS for 40 minutes at 37°C in shaking water path at 100 r.p.m. Cell suspensions obtained will be filtered, then the pellet after centrifugation will be treated with red blood cells lysing solution and washed with PBS.

SUMMARY:
Miscarriage is the most frequently encountered complication of pregnancy ranging from 10% to 30%. The etiology of recurrent spontaneous miscarriage (RSM) in 40%-50% of cases cannot be identified. Immunological disturbances have been suggested to play an important role.

Previous studies have focused that women with miscarriage have elevated NK cell numbers and activity both in the periphery and in the endometrium. Also, NK cells in women with RSM displayed an imbalance of Killer cell Ig-like receptors (KIRs) in favor of activating KIR leading to an unbalanced activation of dNK cytotoxicity and higher risk of miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Regular marital life with the same partner.
* Regularly menstruating before current pregnancy.
* Spontaneous conception.

Exclusion Criteria:

* Women with Polycystic ovarian syndrome or any endocrinal abnormalities like DM, thyroid disorders.
* History of abnormal uterine cavity proved by sonohysterography or hysteroscopy before pregnancy.
* Women with positive consanguinity.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women presented with spontaneous miscarriage
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The percentages of MAIT cells and MAIT cells expressing CD56 and CD16 in comparison with NK cells and NKT cells in both blood and decidua | 24 hours
  All markers will be measured by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt